CLINICAL TRIAL: NCT01471275
Title: The Study of TCM in Prevention and Promote of Community-based Diabetes
Brief Title: Chinese Medicine Treatment of Obesity With Type 2 Diabetes, Dyslipidemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Fengmei Lian, Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 368
Record Dates: First submitted 2011-11-14; First posted 2011-11-15 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Type 2 Diabetes Mellitus ;Obesity,High Triglycerides；TCM
Keywords: type 2 diabetes; obesity; hypertriglyceridemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertriglyceridemia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jiangtangtiaozhi decoction (Experimental)
  Interventions: Drug: Jiangtangtiaozhi decoction
- metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 250 mg or 500mg three times a day
  Other Names: Metformin enteric-coated tablets.
  Arms: metformin
Drug: Jiangtangtiaozhi decoction — 15 grams each time, twice a day, with boiled water
  Other Names: a decoction make of 8 herbs
  Arms: Jiangtangtiaozhi decoction

SUMMARY:
With metformin for the control, evaluate the safety and efficacy of Jiangtangtiaozhi decoction in treatment of obesity with type 2 diabetes, dyslipidemia

DETAILED DESCRIPTION:
Waist circumference, body mass index, triglycerides, glycosylated hemoglobin, blood glucose were evaluated; liver function, kidney function, blood, urine, stool, adverse event recording, evaluation of low blood sugar event log security.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent;
2. waistline male ≥ 90cm, female ≥ 80cm;
3. According to the 1999 WHO standards, meet diagnostic criteria for type 2 diabetes onset and untreated patients, after a screening period (diet + exercise therapy 4 weeks) after the fasting plasma glucose ≥ 7.0mmol • L-1, but fasting blood glucose <13.9mmol • L-1, or 2h postprandial blood glucose ≥ 11.1mmol • L-1; and glycated hemoglobin ≥ 7.0%;
4. After a screening period (diet + exercise therapy 4 weeks) after the triglyceride (TG) ≥ 1.7mmol / L, and TG <5.65mmol / L;
5. TCM for the heat of the gastrointestinal;
6. Age 30-65 years old.

Exclusion Criteria:

1. Patients has been used insulin therapy; previously had a continuous period of 3 months or longer treatment of diabetes(including other Chinese and Western medicine, physical therapy, psychological therapy and health food, etc.) ; enrolled within 1 month before the use of blood glucose and lipids drug treatment;
2. Patients with diabetic complications; or a serious heart, lung, liver, kidney, brain and other serious complications or associated with other primary diseases;
3. Patients with uncontrolled blood pressure control, the systolic blood pressure ≥ 160mmHg or (and) diastolic blood pressure ≥ 100mmHg persons;
4. Patients have diabetic ketoacidosis in the last month, diabetic ketoacidosis and severe infections;
5. Patients with mental illness;
6. Pregnancy, pregnancy or breast-feeding women to prepare;
7. Patients with Chinese medicine allergies; and allergy;
8. Patients with had participated in this study within 1 month have participated or are participating in other clinical studies;
9. In the past five years, patients with alcohol and / or psychoactive substances, drug abuse and dependence;
10. According to the researchers to determine, with the possibility of lower income group or the other into a complex set of diseases or conditions, such as work environment, frequent changes in unstable living environment, the situation could easily lead to lost;
11. Patients taking the dose and type of antihypertensive drugs can not remain stable;
12. Patients taking drugs that affect the quality of the body or health food.
13. Patients with liver, impaired renal function (ALT, AST greater than 2 times the upper limit of normal; serum creatinine greater than the upper limit of normal);
14. Patients are known to lower blood sugar for those who are asymptomatic.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin | 12 weeks

SECONDARY OUTCOMES:
Waistline | 4 weeks
Triglycerides | 12 weeks
Liver function | 4 weeks
Renal function | 4 weeks
Whole blood cell analysis | 4 weeks
Urinalysis | 12 weeks
Adverse events recorded | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Tong, Study Chair — China academy of Chinese medical science
Locations (8):
- China (8):
  - Guang'anmen Hospital of China Academy ofChinese Medical Sciences, Beijing, Beijing Municipality
  - Baoding Hospital of TCM, Baoding, Hebei
  - Affiliated Hospital of Changchun University of TCM, Changchun, Jilin
  - Qinghai Provence Hospital of TCM, Xining, Qinghai
  - Tianjin Dagang Hospital, Dagang, Tianjin Municipality
  - Tianjin University of Traditional Chinese Medicine, First Affiliated Hospital, Tianjin, Tianjin Municipality
  - Yichang City Yiling Hospital, Yichang, Yichang
  - Hangzhou Hospital of TCM, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Yu X, Xu L, Zhou Q, Wu S, Tian J, Piao C, Guo H, Zhang J, Li L, Wu S, Guo M, Hong Y, Pu W, Zhao X, Liu Y, Pang B, Peng Z, Wang S, Lian F, Tong X. The Efficacy and Safety of the Chinese Herbal Formula, JTTZ, for the Treatment of Type 2 Diabetes with Obesity and Hyperlipidemia: A Multicenter Randomized, Positive-Controlled, Open-Label Clinical Trial. Int J Endocrinol. 2018 Apr 1;2018:9519231. doi: 10.1155/2018/9519231. eCollection 2018. PMID 29808092